CLINICAL TRIAL: NCT03813446
Title: A Study to Evaluate the Effectiveness of a Novel Device, the RhythmPadBP, in Accurately Detecting Heart Rhythm and Recording Blood Pressure Simultaneously
Brief Title: Detection of Heart Rhythm and BP With RhythmPadBP
Acronym: SLAF-BP
Status: Completed | Type: Observational
Sponsor: Cardiocity Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016RAK01
Record Dates: First submitted 2017-01-16; First posted 2019-01-23 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Device: RhythmPadBP — Detection of heart rhythm and measurement of blood pressure
  Intervention:
  Patients will start by wearing a consumer SmartWatch (Huwaei SmartWatch 2, which has a CE mark) and a 60 second reading of their wrist Photoplethysmyograph (PPG) will be recorded. This will enable us to compare the PPG from the wrist with the fingertip data collected from the RhythmPadBP.
  The watch will be cleaned with alcohol wipe in the same manner that the RhythmPadBP is cleaned between subjects use.
  Patients will be asked to place their palms of both hands on RhythmPadBP and then the underlying heart rhythm and BP will be recorded. 12-lead ECG and BP reading will be obtained by standard devices for comparison.

SUMMARY:
This study will assess a new device, the RhythmPadBP, which detects heart rhythm and measure blood pressure simply by placing palms of the hands on a pad containing titanium electrodes.

DETAILED DESCRIPTION:
Normally the way a doctor will assess the rhythm of the heart involves asking for an electrocardiogram (ECG) which involves having to remove clothing, and sometimes shaving hair. 10 different leads are attached to stickers that are placed on the chest, and other parts of the body. This is known as a 12-lead ECG and is the standard way that heart-rhythm problems are first investigated. The usual method of measuring blood pressure (BP) involves wrapping a cuff around the arm and inflating it to enough to measure the BP. The reading is then displayed on a monitor. This can sometimes be uncomfortable and is often time consuming, particularly in busy clinical settings.

Recent advances in technology however have given us different ways of gaining some of the same information given by a 12 lead ECG and the standard BP apparatus, using much easier to use devices. One of these devices is the RhythmPadBP system by Cardiocity TM. This is a device where participants can record the underlying heart rhythm and BP readings simply by placing palms of both hands on the device. This device does not require removal of clothing or placing a BP cuff around arm and so the readings can be gained more rapidly and with greater convenience.

Investigators propose to test this device to assess how accurately it recognises the most common cardiac rhythm disturbances, e.g. atrial fibrillation (AF), and also measures the blood pressure. This will help to identify AF and any difference of BP in both arms.

AF is an independent risk factor for stroke and increases the risk of stroke by five-fold. A discrepancy of BP in both arms can be a sign of blood vessel disease and is linked to increased risk of cardiovascular and cerebrovascular disease. If investigators find that this device is correctly recording AF and BP, it may give us another simpler way of diagnosing AF and BP discrepancies on both sides.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater or equal to 18 years
2. Able to consent
3. No known allergies to the metal or any component used in the RhythmPadBP

Exclusion Criteria:

1. Age less than 18 years
2. Not able to consent
3. Allergies to the metal or any component of the RhythmPadBP device
4. Active skin conditions affecting the hands, i.e. burns, infections
5. In-situ cardiac devices i.e. pacemaker or a defibrillator that could interfere with the ECG recording.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending for routine 12-lead ECG, referred by the primary care physician and also patients attending cardiology department at Ashford & St Peters Hospitals NHS Foundation Trust, Chertsey
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Atrial Fibrillation | 18 months
  The diagnosis of Atrial Fibrillation will be achieved through Cardiologist review of p-waves and QRS complexes on both a 1 lead and a 12 lead ECG conducted at the time of study for each participant.

SECONDARY OUTCOMES:
Measurement of BP in both arms with standard BP apparatus Vs RhythmPad BP recordings | 18 months
  Measurement of blood pressure simultaneously from both arms comparing the two procedures. Both systolic and diastolic blood pressure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Riyaz A Kaba, MBBS, FRCP, Principal Investigator — Ashford and St Peter's Hospitals NHS Foundation Trust
Locations (1):
- Ashford and St Peters NHS Trust, Chertsey, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided